CLINICAL TRIAL: NCT05753436
Title: Evaluation of the Effect of Curcumin Administration on the Clinical Outcome of Diabetic Patients With Atherosclerotic Cardiovascular Risk
Brief Title: Curcumin's Effect on Diabetic Patients With Atherosclerotic Cardiovascular Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omar El Rakabawy, Teaching Assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC#120
Record Dates: First submitted 2023-01-31; First posted 2023-03-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Dyslipidemias; Hypertension
Keywords: Diabetes Mellitus; ASCVD Risk; Curcumin; Inflammation; Oxidative stress; Diabetes complication
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias; Hypertension; Diabetes Mellitus; Inflammation; Diabetes Complications | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1, Curcumin group (Active Comparator): Group 1, Curcumin group (n=36): Patients will receive conventional treatment co-administrated with Turmeric Curcumin 500 mg thrice daily for 14 weeks.
  Interventions: Dietary Supplement: Puritans Pride Turmeric curcumin® 500 mg
- Group 2, Control group (No Intervention): Group 2, Control group (n= 36): Patients will receive conventional therapy alone for 14 weeks.

INTERVENTIONS:
Dietary Supplement: Puritans Pride Turmeric curcumin® 500 mg — Turmeric curcumin 500 mg per oral capsule of Puritans Pride company supplement composed of Turmeric (curcuma longa) root 450mg and Turmeric extract (curcuma longa root 50mg ) standardized to contain 95%curcuminoids.It is added because of its possibility to reduce the risk of ASCVD by lowering blood pressure, lipid profile, blood glucose, inflammation, and oxidative stress.
  Other Names: Curcumin
  Arms: Group 1, Curcumin group

SUMMARY:
The aim of the study is to assess the safety and efficacy of Curcumin supplementation in combination to the conventional therapy in improving the clinical outcomes, oxidative stress and inflammation in diabetic patients with risk of ASCVD.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is one of the most devastating consequences of Diabetes Mellitus (DM), especially when combined with other comorbid conditions such as dyslipidemia and hypertension. To lessen the probability of ASCVD, modifying an individual's lifestyle and regulating one's lipid profile, blood pressure, and glucose levels are all beneficial approaches that decrease the risk of ASCVD occurrence. Numerous diseases, including hypertension, dyslipidemia, and diabetes mellitus, have been shown to be significantly influenced by both oxidative stress and inflammation. Curcumin is thought to regulate blood pressure, lipid profile, blood glucose levels. Moreover, It is claimed that curcumin can alleviate inflammation and oxidative stress. Curcumin is therefore suggested to have a beneficial role in lowering the risk of atherosclerotic cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Male or female patients aged 40 years or older
2. A calculated 10 year ASCVD risk score of 5 % or more
3. Patient previously or newly diagnosed with hypertension
4. Patient previously or newly diagnosed with dyslipidaemia
5. Patients diagnosed as Type 2 diabetes mellitus taking insulin or oral hypoglycemic agent with controlled HbA1c < 10%
6. Willingness and ability to give informed consent.

Exclusion Criteria:

1. Congenital or acquired bleeding disorders.
2. Cholelithiasis, gall bladder or biliary tract disease or other active liver diseases.
3. Pregnant or breastfeeding women.
4. Oral hypoglycemic drugs that affect cardiovascular diseases risk.
5. Patients with clinical ASCVD (myocardial infarction, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack, or peripheral arterial disease).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
(Atherosclerotic cardiovascular diseases risk score) Low-risk (<5%) Borderline risk (5% to 7.4%) Intermediate risk (7.5% to 19.9%) High risk (≥20%) | Change from Baseline ASCVD risk scoring at 14 weeks
  10 year ASCVD risk calculation by using Pooled cohort equations
Blood Glucose Level | Change from Baseline Blood Glucose Level at 14 weeks
  Fasting blood glucose (FBG) in mg/dl , Hemoglobin A1c (HbA1c) in percentage
Lipid Profile | Change from Baseline Lipid profile at 14 weeks
  Serum sample to determine ( Triglyceride level , LDL ,HDL ,Total cholesterol ) in mg/dl
Blood Pressure | Change from Baseline Blood Pressure at 14 weeks
  (SBP and DBP) in mmHg by using Sphygmomanometer
Heart Rate | Change from Baseline Heart Rate at 14 weeks
  Pulse in bpm

SECONDARY OUTCOMES:
Concentration of Tumor necrosis factor alpha ( TNF-alpha) | Change from Baseline TNF-alpha concentration at 14 weeks
  Serum sample to determine TNF alpha (Inflammatory biomarker)
Concentration of Malondialdehyde (MDA) | Change from Baseline MDA concentration at 14 weeks
  Serum sample to determine MDA (Oxidative stress marker)
International normalized ratio | Change from Baseline INR level at 14 weeks
  Blood sample to determine INR level for those patients receiving anticoagulants
Serum Ferritin | Change from Baseline Ferritin concentration at 14 weeks
  Serum Ferritin for those patients who are suspected to be anemic or are anemic.

CONTACTS AND LOCATIONS:
Locations (1):
- Demerdash Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No